CLINICAL TRIAL: NCT02762383
Title: A Pilot, Open-Label, Multicentre Study Evaluating the Long-Term Safety and Tolerability of a Low-Dose Peginterferon Alfa-2a Maintenance Monotherapy in Chronic Hepatitis C Patients Co-Infected With Human Immunodeficiency Virus and Who Do Not Respond to a Standard Regimen of Peginterferon Alfa-2a Plus Ribavirin
Brief Title: Pegasys Long-Term Anti-Fibrotic Effect Co-Infection Trial (PERFECT)
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Low recruitment
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ML18234; 2004-002736-26 (EudraCT Number)
Record Dates: First submitted 2016-05-03; First posted 2016-05-04 (Estimated); Last update posted 2016-09-07 (Estimated); Status verified 2016-05

CONDITIONS: HIV/HCV Coinfection
MeSH Terms: interventions — peginterferon alfa-2a

ARMS (1):
- Peginterferon Alfa-2a (Experimental): Participants will receive a low dose of peginterferon alfa-2a for 18 months.
  Interventions: Drug: Peginterferon Alfa-2

INTERVENTIONS:
Drug: Peginterferon Alfa-2 — Peginterferon alfa-2a will be administered as 90 micrograms (mcg) via subcutaneous (SC) injection once weekly.
  Other Names: Pegasys

SUMMARY:
This is an uncontrolled, open-label, Phase III trial of peginterferon alfa-2a (Pegasys) in participants coinfected with human immunodeficiency virus (HIV) and hepatitis C virus (HCV). Participants with HIV/HCV who do not show negative or reduced HCV ribonucleic acid (RNA) after at least 12 weeks of treatment with peginterferon alfa-2a plus ribavirin will receive a low dose of peginterferon alfa-2a for 18 months. The primary objective is to evaluate safety and tolerability. Secondary objectives are to evaluate histological, virological, and biochemical effects.

ELIGIBILITY:
Inclusion Criteria:

* Serologic evidence of chronic hepatitis C infection by anti-HCV antibody test
* Received peginterferon alfa-2a for at least 12 weeks and either did not reach a 2-log drop in HCV RNA after 12 weeks of treatment, did not reach an undetectable HCV RNA after 24 weeks of treatment, or reached undetectable HCV RNA that was detectable again at the end of 48 weeks of treatment
* Detectable serum HCV RNA at Screening
* Serologic evidence of HIV infection by HIV RNA detection
* CD4 cell count greater than or equal to (>/=) 100 cells/mcL during therapy with peginterferon alfa-2a plus ribavirin for at least 12 weeks
* Stable HIV status and, if on antiretroviral therapy, a stable regimen for at least 6 weeks prior to Baseline
* Compensated liver disease
* No evidence of hepatocellular carcinoma

Exclusion Criteria:

* Pregnant or breastfeeding
* Antineoplastic or immunomodulatory treatment within 6 months prior to first dose
* Any investigational drug within 6 weeks prior to first dose
* Positive for hepatitis A immunoglobulin M antibody
* Severe neutropenia or thrombocytopenia at Screening while still on therapy with peginterferon alfa-2a plus ribavirin
* Severe psychiatric or neurologic comorbidity
* History of any significant medical conditions, such as immune disorders or disease of the major organ systems
* Uncontrolled thyroid disease
* Severe retinopathy
* Evidence of drug abuse

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2005-03; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants with Adverse Events (AEs) | From Baseline to end of treatment (up to 18 months)

SECONDARY OUTCOMES:
Percentage of Participants with Histological Response According to Paired Biopsy | At end of treatment (up to 18 months)
HIV RNA Viral Load in Copies per Milliliter (copies/mL) | At end of treatment (up to 18 months)
Cluster of Differentiation (CD) 4 Cell Count in Cells per Microliter (cells/mcL) | At end of treatment (up to 18 months)
Percentage of Participants with Virological Response According to HCV RNA Viral Load | At 6, 12, and 18 months during treatment, and at 24 weeks after end of treatment (up to 2 years overall)
Percentage of Participants with Biochemical Response According to Alanine Aminotransferase (ALT) Level | At end of treatment (up to 18 months)
Percentage of Participants with Sustained Biochemical Response According to ALT Level | At 24 weeks after end of treatment (up to 2 years overall)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Chair — Hoffmann-La Roche
Locations (6):
- Belgium (6):
  - Brussels
  - Charleroi
  - Edegem
  - Ghent
  - Leuven
  - Liège